CLINICAL TRIAL: NCT05854368
Title: Circulating Biomarker Signatures for the Detection of Gastric Preneoplasia and Cancer
Acronym: PREGASIGN#1
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Pasteur (Industry)
Collaborators: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2021-097
Record Dates: First submitted 2023-02-08; First posted 2023-05-11 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Gastric Lesion; Gastric Precancerous Condition; Gastric Cancer
Keywords: Gastric Cancer, biomarkers,
MeSH Terms: conditions — Stomach Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: Patients with gastric lesion (including preneoplasia or cancer) and Healthy Volunteers (control)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with gastric lesion (Other): Patients with:
  * Gastric epithelial dysplasia
  * Glandular atrophy of the gastric mucosa
  * Intestinal metaplasia of the gastric mucosa
  * Proximal gastric adenocarcinoma
  * Distal gastric adenocarcinoma
  Interventions: Procedure: Additional blood collection as part of a blood sampling performed during routine care or specific for the research if not part of routine care.
- Control (Other): Healthy Volunteers
  Interventions: Procedure: Blood collection

INTERVENTIONS:
Procedure: Additional blood collection as part of a blood sampling performed during routine care or specific for the research if not part of routine care. — Collection of an additional blood volume (9 mL) as part of a blood sampling performed during routine care or specific for the research if not part of routine care.
  Arms: Patients with gastric lesion
Procedure: Blood collection — Blood sample collection (10 mL)
  Arms: Control

SUMMARY:
The goal of this study is to characterize and validate a signature of circulating biomarkers in plasma, associated with the presence of gastric preneoplasia in patients with preexisting gastric lesion compared with a control group.

For this purpose:

* Patients with pre-existing gastric lesions will be invited to participate to this study. If they are willing to participate an additional blood sample (9 mL) will be collected at the time of the blood collection performed during their routine care
* Healthy subjects will be invited to participate to constitute the control group. If they are willing to participate a blood sample (9 ml) will be drawn specifically for this study

DETAILED DESCRIPTION:
Gastric cancer (GC) is the fourth cause of cancer-related death and the fifth most common diagnosed cancer worldwide with 1 million new cases per year. GC is mainly associated with a poor prognosis, highlighting the importance of its early detection. GC results from a multistep process starting from a gastric chronic inflammation preceding atrophic gastritis (AG), the development of preneoplasia (intestinal metaplasia (IM), dysplasia (Dys) and then cancer lesions. Presently, GC can only be diagnosed by endoscopy, which is an invasive, and costly method with its limits. Indeed, preneoplasia as Dys can escape endoscopic detection. Therefore, the discovery of blood-based biomarkers to identify the presence of gastric preneoplasia and/or cancer lesions at the earliest, at an asymptomatic stage, is of paramount interest. It is crucial not only for the early detection/prevention of individuals at risk of GC but also useful for patient follow-up to predict disease recurrence/outcome and to monitor treatment. Using plasma samples from patients at various stages of the GC cascade, we previously identified two signatures of 6 protein candidates to predict the presence of preneoplasia and GC lesions. Based on these data, the goal of this study is to further test and validate these different signatures, and to improve their predictive ability at the earliest stages of the GC cascade, taking into account the different types of gastric preneoplasia, IM and Dys, and their grade of severity. To achieve this goal, a large multicentric cohort of patients will be established including different groups of plasma samples covering the most complete panel of the type/grades of gastric preneoplasia as well as at early stages of GC. These plasma samples will be then used to measure the level of the different signature components using various method of analysis as immuno-based assays.

ELIGIBILITY:
Inclusion Criteria:

Common

* 18 years old or highter
* written informed consent prior to any study procedure
* Affiliated to a social insurance system

Specific to patients with gastric lesions

* Untreated glandular atrophy (with or without intestinal metaplasia and/or dysplasia) and histologically diagnosed as of 2014
* Treatment naïve Gastric cancer (distal or proximal adenocarcinoma)

Exclusion Criteria:

Common

* Autoimmune disease or disease that impacts the immune system (e.g: HIV)
* Chronic inflammatory disease
* Known evolutive cancer (excluding gastric cancer)
* Treated in the last 3 months or currently treated with therapy that interferes with the immune system (e.g. immunosuppressive therapy)
* Current treatment with long-term corticosteroid therapy
* Current treatment with long-term nonsteroidal anti-inflammatory drugs
* Pregnant woman or breastfeeding
* Patient or healthy volunteer under legal protection (e.g. guardianship)
* Patient or healthy volunteer currently participating to a clinical trial evaluating either an experimental medical product or a medical device
* Patient or healthy volunteer currently in custody

Specific to Healthy Volunteer

* Known history of Helicobacter pylori infection
* Known history of gastric lesions (i.e. chronic gastritis, gastric atrophy, intestinal metaplasia, dysplasia and cancer)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2500 (Estimated)
Dates: Start 2023-07-03 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Characterization and validation of a signature combining plasmatic proteins related to inflammation and carcinogenesis process, associated with the presence of gastric mucosal dysplasia lesions compared with an H. pylori negative control group. | 30 months
  From the plasma obtained from patients previously diagnosed by gastric endoscopy for the presence of dysplasia in the gastric mucosa and that have signed a prior consent form, the concentration of protein biomarker candidates will be determined using a bead-based immunoassay according to Luminex® technology. It will be expressed as amount per ml of plasma. For each protein constituting the signature of biomarkers, its levels in the plasma of patients with dysplasia will be compared to the corresponding levels in healthy subjects with a negative H. pylori serology and referred as a control group.

SECONDARY OUTCOMES:
Characterization and validation of a signature combining plasmatic proteins related to inflammation and carcinogenesis process, associated with the presence of glandular atrophy lesions compared with an H. pylori negative control group. | 30 months
  From the plasma obtained from patients previously diagnosed by gastric endoscopy for the presence of glandular atrophy lesions in the gastric mucosa and that have signed a prior consent form, the concentration of protein biomarker candidates will be determined using a bead-based immunoassay according to Luminex® technology. It will be expressed as amount per ml of plasma. For each protein constituting the signature of biomarkers , its levels in the plasma of patients with gastric glandular atrophy lesions will be compared to the corresponding levels in healthy subjects with a negative H. pylori serology and referred as a control group.
Characterization and validation of a signature combining plasmatic proteins related to inflammation and carcinogenesis process, associated with the presence of intestinal metaplastic lesions compared with an H. pylori negative control group. | 30 months
  From the plasma obtained from patients previously diagnosed by gastric endoscopy for the presence of intestinal metaplastic lesions within the gastric mucosa and that have signed a prior consent form, the concentration of protein biomarker candidates will be determined using a bead-based immunoassay according to Luminex® technology. It will be expressed as amount per ml of plasma. For each protein constituting the signature of biomarkers, its levels in the plasma of patients with gastric intestinal metaplastic lesions will be compared to the corresponding levels in healthy subjects with a negative H. pylori serology and referred as a control group.
Characterization and validation of a signature combining plasmatic proteins related to inflammation and carcinogenesis process, associated with the presence of proximal gastric adenocarcinoma compared with an H. pylori negative control group. | 30 months
  From the plasma obtained from patients previously diagnosed by gastric endoscopy for the presence of proximal gastric adenocarcinoma and that have signed a prior consent form, the concentration of protein biomarker candidates will be determined using a bead-based immunoassay according to Luminex® technology. It will be expressed as amount per ml of plasma. For each protein constituting the signature of biomarkers, its levels in the plasma of patients with proximal gastric adenocarcinoma will be compared to the corresponding levels in healthy subjects with a negative H. pylori serology and referred as a control group.
Characterization and validation of a signature combining plasmatic proteins related to inflammation and carcinogenesis process, associated with the presence of distal gastric adenocarcinoma compared with an H. pylori negative control group. | 30 months
  From the plasma obtained from patients previously diagnosed by gastric endoscopy for the presence of distal gastric adenocarcinoma and that have signed a prior consent form, the concentration of protein biomarker candidates will be determined using a bead-based immunoassay according to Luminex® technology. It will be expressed as amount per ml of plasma. For each protein constituting the signature of biomarkers, its levels in the plasma of patients with distal gastric adenocarcinoma will be compared to the corresponding levels in healthy subjects with a negative H. pylori serology and referred as a control group.
Characterization of the plasma levels of the proteins biomarker composing these signatures specific for the different stages of gastric cancer cascade, between the different studied pathology groups | 30 months
  From the plasma obtained from patients previously diagnosed by gastric endoscopy for the presence of gastric lesions at the different stages of the gastric cancer cascade (dysplasia, glandular atrophy, intestinal metaplasia, proximal gastric adenocarcinoma and distal gastric adenocarcinoma), and that have signed a prior consent form, the concentration of protein biomarker candidates will be determined using a bead-based immunoassay according to Luminex® technology. It will be expressed as amount per ml of plasma. For each protein constituting the signature of biomarkers , its plasma levels will be compared between patients from the different groups of gastric lesions dysplasia, glandular atrophy, intestinal metaplasia, proximal gastric adenocarcinoma and distal gastric adenocarcinoma).

CONTACTS AND LOCATIONS:
Overall Officials: Dominique LAMARQUE, MD, PhD, Principal Investigator — Ambroise Paré Teaching Hospital (AP-HP)
Locations (7):
- France (7):
  - Ambroise Paré Teaching Hospital (AP-HP), Boulogne-Billancourt
  - Beaujon Teaching Hospital (AP-HP), Clichy
  - Kremlin Bicêtre Teaching Hospital (AP-HP), Le Kremlin-Bicêtre
  - Cochin Teaching Hospital (AP-HP), Paris
  - INVOLvE - Investigation et volontaires en santé humaine (Institut Pasteur), Paris
  - Saint Antoine Teaching Hospital (AP-HP), Paris
  - Saint Louis Teaching Hospital (AP-HP), Paris

REFERENCES:
- [Background] Kotilea K, Bontems P, Touati E. Epidemiology, Diagnosis and Risk Factors of Helicobacter pylori Infection. Adv Exp Med Biol. 2019;1149:17-33. doi: 10.1007/5584_2019_357. PMID 31016621